CLINICAL TRIAL: NCT01022762
Title: A 16-week, Multicentre, Randomised, Open-label, Parallel Group Study to Investigate the Efficacy and Safety Profiles of Repaglinide Monotherapy Compared to Gliclazide Monotherapy in Chinese Antidiabetic-naïve Subjects With Type 2 Diabetes
Brief Title: Comparison of Repaglinide and Gliclazide in Chinese Subjects With Type 2 Diabetes Never Received Oral Antidiabetic Drug Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGEE-3783; U1111-1111-9453 (Other: WHO)
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Results first posted 2011-12-29 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; Gliclazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- repaglinide (Active Comparator): 1 mg repaglinide twice daily (weeks 0-4), titrated (individually adjusted) to maintenance dose (weeks 4-16). Maximum dose is 4 mg three times daily
  Interventions: Drug: repaglinide
- gliclazide (Active Comparator): 80 mg gliclazide once daily (weeks 0-4), titrated (individually adjusted) to maintenance dose (weeks 4-16). Maximum dose is 160 mg twice daily
  Interventions: Drug: gliclazide

INTERVENTIONS:
Drug: repaglinide — Individually adjusted dose for 16 weeks
  Arms: repaglinide
Drug: gliclazide — Individually adjusted dose for 16 weeks
  Arms: gliclazide

SUMMARY:
This trial is conducted in Asia. The aim of this clinical trial is to investigate the blood glucose lowering effect and the safety profile of repaglinide given alone compared to gliclazide given alone in Chinese subjects with type 2 diabetes who never have been treated with oral anti-diabetic drugs (OADs). This study also investigates the augment effect of repaglinide on the phases of insulin secretion as a subgroup study.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Oral anti-diabetic drug (OAD) naïve (unsystematic OAD treatment 6 months prior to this trial is allowed)
* Insulin naïve (less than 1 week of daily use of insulin therapy before trial start is allowed)
* Lipid-lowing agent naïve
* HbA1c: 6.5-8.5%
* Fasting glucose: 6.1-13.0 mmol/L (110-234 mg/dl)
* Body Mass Index (BMI): 20-35 kg/m^2
* Be able and willing to perform self-monitored plasma glucose (SMPG)
* Be able and willing to eat 3 main meals per day
* Only applicable to subjects who will participate in the subgroup study: Be able and willing to perform and complete IVGTT (intravenous glucose tolerance test) at additional visits

Exclusion Criteria:

* Known or suspected allergy to repaglinide, gliclazide, or related products (for example sulfonamide or other sulphonylureas (SUs)), or any of the excipients in the study drugs
* Previous participation in this study
* Participation in a study of another investigational drug within 1 month prior to study start

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Shanghai, Shanghai Municipality, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 23 sites in China.
Pre-assignment Details: Between screening and treatment with trial drug the participants were assessed for eligibility and were randomised to one of two treatment arms. A sub-group of 69 participants was recruited for intravenous glucose tolerance test and randomised into the repaglinide treatment group (35 participants) and gliclazide treatment group (34 participants)
Period: Overall Study
Arm/Group | Repaglinide | Gliclazide
Started | 218 | 222
Exposed to Trial Drug | 217 (One participant was not exposed to the treatment due to fulfillment of exclusion criteria) | 218 (Four participants were not exposed to the treatment due to non-compliance or lost to follow-up)
Completed | 196 | 194
Not Completed | 22 | 28
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 7 | 6
Not completed — Unclassified | 12 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Repaglinide | Gliclazide | Total
Number analyzed (Participants) | 217 | 218 | 435
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (10.0) | 53.5 (9.9) | 53.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 95 | 202
  Male | 110 | 123 | 233
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 217 | 218 | 435
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 217 | 218 | 435
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 217 | 218 | 435
Height [Mean (Standard Deviation); unit: cm] | 163.2 (8.9) | 163.9 (8.4) | 163.5 (8.7)
Weight [Mean (Standard Deviation); unit: kg] | 68.7 (11.6) | 68.4 (11.2) | 68.6 (11.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.69 (3.00) | 25.37 (3.01) | 25.53 (3.00)
Duration of diagnosed diabetes [Mean (Standard Deviation); unit: years] | 1.02 (1.95) | 0.79 (1.82) | 0.91 (1.89)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Time Frame: Week 0, week 16
Population: Full analysis set (FAS) is randomised participants exposed to at least one dose of trial product after randomisation. Missing values were replaced with the last post-baseline data based on LOCF (last observation carried forward).
Measure: Least Squares Mean (Standard Error); unit: percentage (%) of total haemoglobin
Arm/Group | Repaglinide | Gliclazide
Number analyzed (Participants) | 206 | 202
percentage (%) of total haemoglobin | -0.857 (0.051) | -0.871 (0.051)
Statistical Analysis 1: Comparison: Repaglinide vs Gliclazide; H0: Change from baseline in HbA1c of repaglinide therapy at 16 weeks of treatment - change from baseline in HbA1c of gliclazide therapy at 16 weeks of treatment >= 0.4%. H1: Change from baseline in HbA1c of repaglinide therapy at 16 weeks of treatment - change from baseline in HbA1c of gliclazide therapy at 16 weeks of treatment < 0.4%. Sample size was calculated to achieve a power of at least 85%, assuming an equal change in HbA1c and a common standard deviation of 1.2%; Test type: Non-Inferiority or Equivalence — Non-inferiority would be shown if the upper limit of the 95% confidence interval was less than 0.4%. This corresponds to a one-sided test with a significance level of 2.5% of the hypothesis; ANCOVA — The p-value corresponds to one-sided hypotheses of superiority with a significance level of 2.5%; ANCOVA model was with treatment, centre as explanatory variables and baseline HbA1c value as covariate; Mean Difference (Net) = 0.014, 95% CI [-0.115 to 0.143], Standard Error of Mean 0.066 — If non-inferiority of repaglinide alone was shown, a test for superiority would be performed based on FAS. Superiority of repaglinide alone over gliclazide alone would be claimed if the upper limit of the 95% CI for the difference was lower than 0%

2. Secondary Outcome: Change in Fasting Plasma Glucose
Time Frame: Week 0, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Repaglinide | Gliclazide
Number analyzed (Participants) | 203 | 200
mmol/L | -1.409 (0.104) | -1.667 (0.102)

3. Secondary Outcome: Change in 2-hour Postprandial Plasma Glucose (PPG) Over a Standard Meal
Description: A standard meal contains 100g carbohydrate
Time Frame: Week 0, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Repaglinide | Gliclazide
Number analyzed (Participants) | 203 | 199
mmol/L | -0.596 (0.215) | -0.699 (0.211)

4. Secondary Outcome: Percentage of Participants Achieving the Treatment Target of HbA1c Below or Equal to 6.5%
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Repaglinide | Gliclazide
Number analyzed (Participants) | 217 | 218
percentage of participants | 62 | 59

5. Secondary Outcome: Change in Fasting Serum Free Fatty Acid (FFA) From Baseline
Time Frame: Week 0, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Repaglinide | Gliclazide
Number analyzed (Participants) | 206 | 202
mmol/L | -0.012 (0.014) | -0.02 (0.014)

6. Secondary Outcome: Change in 2-hour Postprandial Serum Free Fatty Acid (FFA) Over a Standard Meal
Time Frame: Week 0, week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Repaglinide | Gliclazide
Number analyzed (Participants) | 204 | 201
mmol/L | -0.003 (0.007) | -0.004 (0.007)

7. Secondary Outcome: Change in AUC0-180 of Serum Insulin Concentration of IVGTT (Intravenous Glucose Tolerance Test)
Time Frame: Over the course of three hours at Week 0 and Week 16
Population: A total of 69 participants were recruited into IVGTT, and were randomised into repaglinide treatment group (35 participants) and gliclazide treatment group (34 participants). Participants with eligible IVGTT profiles were included in IVGTT analysis set.
Measure: Mean (Standard Deviation); unit: min*pmol/L
Arm/Group | Repaglinide | Gliclazide
Number analyzed (Participants) | 31 | 31
min*pmol/L | 5139.55 (8720.80) | 1426.21 (5262.15)

8. Secondary Outcome: Change in AUC0-180 of Plasma Glucose Concentration of IVGTT
Time Frame: Over the course of three hours at Week 0 and Week 16
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: min*mmol/L
Arm/Group | Repaglinide | Gliclazide
Number analyzed (Participants) | 31 | 31
min*mmol/L | -272.30 (290.79) | -348.03 (258.86)

9. Secondary Outcome: Number of All Treatment Emergent Hypoglycaemic Episodes
Description: A hypoglycaemic episode was defined as treatment emergent if the onset of the episode was on or after the first day of trial product and no later than the last day of the trial product.
Time Frame: Weeks 0-16
Population: Safety analysis set contains all randomised participants exposed to at least one dose of trial drug(s). One participant was randomised into repaglinide group, but was dispensed gliclazide from the very beginning of the study due to the investigator's negligence. This participant continued the gliclazide treatment until the end of the study.
Measure: Number; unit: episodes
Arm/Group | Repaglinide | Gliclazide
Number analyzed (Participants) | 216 | 219
episodes | 165 | 147

10. Secondary Outcome: Cholesterol
Description: The number of participants having a change in cholesterol from "normal" to "abnormal". "Abnormal" means a value of blood cholesterol is out of the normal range.
Time Frame: Week 0, week 16
Population: Safety analysis set contains all randomised participants exposed to at least one dose of trial drug(s)
Measure: Number; unit: participants
Arm/Group | Repaglinide | Gliclazide
Number analyzed (Participants) | 216 | 219
participants | 18 | 11

11. Secondary Outcome: Change in Body Weight
Time Frame: Week 0, week 16
Population: Full analysis set (FAS) is randomised participants exposed to at least one dose of trial product after randomisation
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Repaglinide | Gliclazide
Number analyzed (Participants) | 196 | 194
kg | -0.750 (0.218) | -0.511 (0.215)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a timespan of 16 weeks.
Description: Safety analysis set contains all randomised participants exposed to at least one dose of trial drug(s).
Arm/Group | Repaglinide | Gliclazide
Serious Adverse Events (participants affected / at risk) | 3/216 | 0/219
Other Adverse Events (participants affected / at risk) | 0/216 | 0/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Repaglinide (N=216) | Gliclazide (N=219)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gall bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to not release data until specified milestones, e.g. when the clinical trial report is available. This includes the right to not release interim results of clinical trials. At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.